CLINICAL TRIAL: NCT02107482
Title: Bilateral Comparator, Sham-Light Source Controlled, Assessor Blinded Clinical Trial of Localized Narrow Band-Ultraviolet B (NB-UVB) (Levia®) Treatment for Plaque-type Psoriasis
Brief Title: Use of Localized NB-UVB (Levia®) in the Treatment of Plaque-psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Levia
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Results first posted 2017-02-20 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levia Narrow Band UVB (Active Comparator): Levia Narrow Band UVB dosing for subjects with skin type I: starting dose of 195 mj/cm2, for subjects with skin type II: starting dose of 330 mj/cm2, for subjects with skin type III: starting dose of 390 mj/cm2, for subjects with skin type IV: starting dose of 495 mj/cm2, for subjects with skin type V: starting dose of 525 mj/cm2, for subjects with skin type VI: starting dose of 600 mj/cm2. The dose will be increased by 15% with each treatment, as long as there are no side effects with treatment such as burning or redness.
  Interventions: Device: Levia Narrow Band UVB
- Levia sham/visible-light source (Sham Comparator): the light is produced using the same Levia® device. Levia® enable the user to switch off the UVB light and only produce visible light spectrum.
  Interventions: Device: Levia sham/visible-light source

INTERVENTIONS:
Device: Levia Narrow Band UVB — The device's spectral output is is Narrow Band UVB (NB-UVB) (NB-Levia): 308-312 nm
  Arms: Levia Narrow Band UVB
Device: Levia sham/visible-light source — the light spectrum is in the range of 400-700nm, the light is produced using the same Levia® device. Levia® enable the user to switch off the UVB light and only produce visible light spectrum.
  Arms: Levia sham/visible-light source

SUMMARY:
The purpose of the study is to test the effect of a localized narrow band ultraviolet (NB-UVB) phototherapy compared to visible light that does not produce UVB on the clearance of psoriasis plaques and resolution of itching. Localized NB-UVB (Levia®) phototherapy device is cleared by the U.S Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
This will be an ascending dose study with treatments three times per week, initial treatment dose and increasing regimen is adjusted according to the subject skin type. A suggested treatment regimen schedule provided from Lerner Medical Devices, Inc:

For subjects with skin type I: starting dose of 195 mj/cm2, for subjects with skin type II: starting dose of 330 mj/cm2, for subjects with skin type III: starting dose of 390 mj/cm2, for subjects with skin type IV: starting dose of 495 mj/cm2, for subjects with skin type V: starting dose of 525 mj/cm2, for subjects with skin type VI: starting dose of 600 mj/cm2.

The dose will be increased by 15% with each treatment, as long as there are no side effects with treatment such as burning or redness.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older with bilateral psoriasis plaques, in general good health as determined by the Principal Investigator by medical history and physical exam.
* Able to understand consent procedure
* Able to comply with protocol activities
* Must have baseline symmetric target lesions with baseline Target Lesion Score (TLS) of 6 or higher (scale of 0-12), i.e., moderate in intensity for each target.

Target Lesion Scoring: Thickness, scaling and erythema of the plaques are rated each on a scale of 0-4. The three scores are summed. The minimum score is 0; the maximum is 12. Scores of 6 or greater are considered moderate to severe.

Exclusion Criteria:

* Patients less than 18 years old
* Patients not able to understand consent procedure
* Patients unable to comply with protocol activities
* Non-English speakers: the study assessments/questionnaires/evaluations are not scientifically validated in languages other than English
* Baseline target lesions scores of less than 6
* Patients with a photosensitive disorder or on a medication which has been demonstrated in these patients to cause photosensitivity
* Patients receiving concomitant phototherapy to test sites
* Patient receiving topical medication to test sites within 2 weeks of study initiation
* Patient receiving Methotrexate, Acitretin, Cyclosporine, or other oral medications for psoriasis within 4 weeks of study initiation
* Patients receiving Etanercept (Enbrel®) within the past 2 months of study initiation
* Patients receiving Infliximab (Remicade®), Ustekinumab (Stelara®), Golimumab (Simponi®) Adalimumab (Humira®) or Alefacept (Amevive®) within the past 3 months prior to study initiation
* Receipt of an investigation agent within the past 4 weeks (or within 5 half lives) prior to study ignition
* Systemic corticosteroid therapy within the past month
* Concurrent use of prohibited medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice b Gottlieb, MD, PhD, Principal Investigator — Tufts Medical Center
Locations (1):
- Dermatology Research, Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Levin AA, Aleissa S, Dumont N, Martinez F, Donovan C, Au SC, Hasanain A, Gottlieb AB. A randomized, prospective, sham-controlled study of localized narrow-band UVB phototherapy in the treatment of plaque psoriasis. J Drugs Dermatol. 2014 Aug;13(8):922-6. PMID 25116969

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Each subject will have a targeted lesion treated with Levia Narrow Band UVB( skin type I: starting dose of 195 mj/cm2, skin type II: starting dose of 330 mj/cm2, skin type III: starting dose of 390 mj/cm2, skin type IV: starting dose of 495 mj/cm2, skin type V: starting dose of 525 mj/cm2, skin type VI: starting dose of 600 mj/cm2). The dose will be increased by 15% with each treatment, as long as there are no side effects with treatment such as burning or redness. The same subject will have a second target lesion treated with the Sham Comparator.
Period: Overall Study
Arm/Group | All Participants
Started | 21 (21 participants enrolled. Total of 21 participants recvd both active and sham)
Completed | 17
Not Completed | 4
Not completed — inconveinence | 2
Not completed — Lost to Follow-up | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants - Levia Narrow Band UVB: Each subject will have a targeted lesion treated with Levia Narrow Band UVB( skin type I: starting dose of 195 mj/cm2, skin type II: starting dose of 330 mj/cm2, skin type III: starting dose of 390 mj/cm2, skin type IV: starting dose of 495 mj/cm2, skin type V: starting dose of 525 mj/cm2, skin type VI: starting dose of 600 mj/cm2). The dose will be increased by 15% with each treatment, as long as there are no side effects with treatment such as burning or redness. The same subject will have a second target lesion treated with the Sham Comparator.
Arm/Group | All Participants - Levia Narrow Band UVB
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 48.5 [25 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 6
Race/Ethnicity, Customized [Number; unit: participants]
  white | 20
  African american | 1
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Lesions With a Clear or Almost Clear Rating (Target Lesion Score of 3 or Less) on Target Lesion Scoring at Week 12
Time Frame: 12 weeks
Measure: Number; unit: percentage of lesions changed
Arm/Group | All Participants
Number analyzed (Participants) | 21
percentage of lesions changed
  Levia Narrow Band UVB | 47.6
  Levia Sham | 33.3

2. Secondary Outcome: The Percentage of Change in Target Lesion Score
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of change in TLS
Arm/Group | All Participants
Number analyzed (Participants) | 21
percentage of change in TLS
  Levia Narrow Band UVB | 47 (0.8)
  Levia Sham | 29 (0.8)

3. Secondary Outcome: Changes in Target Lesion Pruritus Visual Analog Scale (VAS) at Week 12
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Percent Change in Target Lesion Pruritus
Arm/Group | All Participants
Number analyzed (Participants) | 21
Percent Change in Target Lesion Pruritus
  Levia Narrow baned UVB | 62 (0.8)
  Levia Sham | 27 (0.8)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 8/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=21)
burn (Skin and subcutaneous tissue disorders) | 8 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No